CLINICAL TRIAL: NCT01754896
Title: Pilot Evaluation of Fecal Immunologic Test (FIT) in Ontario
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 209-2011
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; fecal immunochemical test; fecal occult blood test; screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mail-out/Mail-back (Experimental): Mailing of FIT kit directly to patient. Mailing completed kits in for processing.
  Interventions: Other: mailing of FIT kit directly to patient; Other: mailing completed kits in for processing
- Mail-out/Drop-off (Experimental): Mailing of FIT kit directly to patient. Dropping completed kits at lab for processing.
  Interventions: Other: mailing of FIT kit directly to patient; Other: dropping completed kits at lab for processing
- Pick-up/Mail-back (Experimental): Mailed invitation to pick up lab requisition and then kit. Mailing completed kits in for processing.
  Interventions: Other: mailed invitation to pick up lab requisition and then kit; Other: mailing completed kits in for processing
- Pick-up/Drop-off (Experimental): Mailed invitation to pick up lab requisition and then kit. Dropping completed kits at lab for processing.
  Interventions: Other: mailed invitation to pick up lab requisition and then kit; Other: dropping completed kits at lab for processing

INTERVENTIONS:
Other: mailing of FIT kit directly to patient — Patient receives a mailed invitation to participate in CRC screening, with a FIT screening kit included.
  Arms: Mail-out/Drop-off; Mail-out/Mail-back
Other: mailed invitation to pick up lab requisition and then kit — Patients receives a mailed invitation to visit their physician to discuss CRC screening. At that visit, they would receive a FIT laboratory requisition, which they will take to a local lab patient service centre to pick up a FIT kit.
  Arms: Pick-up/Drop-off; Pick-up/Mail-back
Other: mailing completed kits in for processing — Patients mails completed kit in for processing using postage-paid reply envelope provided.
  Arms: Mail-out/Mail-back; Pick-up/Mail-back
Other: dropping completed kits at lab for processing — Patient takes completed FIT in to lab patient service centre for processing.
  Arms: Mail-out/Drop-off; Pick-up/Drop-off

SUMMARY:
Prior to implementation of new colorectal cancer (CRC) screening technology (fecal immunochemical test - FIT) in Ontario, there is a need for a laboratory and field assessment to validate and optimize its use in the Ontario climate and conditions (e.g., large geographic area) and to determine whether adjustments to the current structure of the ColonCancerCheck (CCC) Program would be required.

This study consists of 2 phases. Phase 1 consists of laboratory testing of FIT kits to evaluate analytical performance relevant to the requirements of the CCC Program. Phase 2 is a field assessment to evaluate the effect of different distribution and return methods and pre-labeling of kits on uptake and completion of the tests. The entire study will take 12-18 months to complete, with patients being recruited through family physicians in patient enrollment model (PEM) family practices across the province of Ontario.

This Clinical Trials registration relates to Phase 2 of the study.

DETAILED DESCRIPTION:
In 2008 Ontario launched the ColonCancerCheck (CCC) Program, an organized colorectal cancer (CRC) screening program in which average risk patients are offered an at-home screening test and increased risk patients are offered colonoscopy directly through their family physician.

Currently, Ontario's CCC Program utilizes guaiac fecal occult blood testing (gFOBT) in persons at average risk of CRC. However, the program is currently considering a change to fecal immunochemical testing (FIT).

FIT, which comes in quantitative and qualitative formats, is superior to the gFOBT from a scientific perspective because it specifically detects human hemoglobin. gFOBT uses an indirect detection which depends on a peroxidase reaction not specific for human hemoglobin. FIT methodology is also both more convenient and superior from a participant perspective and multiple studies have demonstrated higher participation rates and improved detection of CRC precursors as well as invasive CRCs with FIT compared to gFOBT.

Organized CRC screening programs considering quantitative FIT face certain additional challenges, including uncertain stability over time and tolerance to variation in temperature following sample collection and prior to arrival in a testing laboratory. Prior to implementation of FIT in Ontario, there is a need for a laboratory and field assessment to validate and optimize its use in the Ontario climate and conditions (e.g., large geographic area) and to determine whether adjustments to the current structure of the CCC Program would be required.

This study consists of 2 phases. Phase 1, laboratory testing, assesses 2 quantitative and 3 qualitative FIT kits to evaluate analytical performance relevant to the requirements of the CCC Program. Phase 2 is a field assessment to evaluate the effect of different distribution and return methods and pre-labeling of kits on uptake and completion of the tests. The entire study will take 12-18 months to complete, with patients being recruited through family physicians in patient enrollment model (PEM) family practices across the province of Ontario. Data collection will take place for 6 months, starting on the day that screening kits and/or invitation letters are mailed to patients.

This Clinical Trials registration relates to Phase 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Physician in Ontario with a patient enrollment model
* patient: 50-74, Ontario resident, enrolled with physician

Exclusion Criteria:

* patient: no personal or first degree relative family history of CRC, no FOBT within prior 5 years, colonoscopy within past 10 years, FOBT within past 2 years

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
FIT Kit uptake | September 2012 to April 2013
  Comparing FIT kit uptake by patients invited to complete fecal occult blood screening for colorectal cancer using a Fecal Immunochemical Test (FIT), and provided with different kit distribution and return methods.

SECONDARY OUTCOMES:
Rejection rates | September 2012 to April 2013
  Assessing the impact of pre-labeling of FIT Kit collection vials with patient name and date of birth, compared to allowing hand-written labeling, on rates of kit rejection at the lab.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Tinmouth, MD, PhD, Principal Investigator — Sunnybrook Research Institute; Linda Rabeneck, MD, MPH, Principal Investigator — Cancer Care Ontario; Lawrence Paszat, MD, SM, Principal Investigator — Institute for Clinical Evaluative Studies (ICES); Nancy Baxter, MD, PhD, Principal Investigator — St. Michaels Hospital; Edward Randall, PhD, DCC, Principal Investigator — Eastern Health
Locations (1):
- Dr. Jill Tinmouth, Toronto, Ontario, Canada